CLINICAL TRIAL: NCT05737459
Title: The Effect of Sedation on Postoperative Cognitive Functions in Patients Operated for Hip Fracture Under Spinal Anesthesia
Brief Title: Sedation and Postoperative Cognitive Functions
Status: Completed | Type: Observational
Sponsor: Izmir Ataturk Training and Research Hospital (Other)
Responsible Party: Principal Investigator, Derya Arslan Yurtlu, Associate Professor, Izmir Ataturk Training and Research Hospital
Other Study IDs: IAERH
Record Dates: First submitted 2023-02-02; First posted 2023-02-21 (Actual); Last update posted 2023-02-21 (Actual); Status verified 2023-02

CONDITIONS: Cognitive Impairment; Femoral Fractures
Keywords: Cognitive Impairment; Mini mental status test; Hip fractures; Ketamine; dexmedetomidine
MeSH Terms: conditions — Cognitive Dysfunction; Femoral Fractures; Hip Fractures

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Days
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Group K: Those who have been administered ketamine for perioperative sedation
- Group D: Those who have been administered dexmedetomidine for perioperative sedation.

SUMMARY:
Patients over the age of 65 who underwent elective surgery for a hip fracture and were sedated during spinal anesthesia were included in the study. Patients who were given ketamine and dexmedetomidine for sedation were included in the study. The Mini Mental Status Tests of the patients measured on the first and third days of the operation in the preoperative period were determined from the hospital records and recorded.

DETAILED DESCRIPTION:
Patients over the age of 65 who underwent elective surgery for a hip fracture and were sedated during spinal anesthesia were included in the study. The cognitive functions of these patients, which were evaluated by a Mini-Mental Test in the preoperative period, on the first and third days of surgery, were recorded from routine patient follow-up forms.

Sedation scores of the patients evaluated by Intraoperative Alertness/Sedation Scale (OAA/S) Observer Evaluation were recorded. Intraoperative hemodynamic data were recorded. The interventions applied to the patient were performed by anesthesiologists who were not involved in the study according to their preferences as part of the routine. The researchers were not involved in any intervention performed on the patient, only the data were recorded.

ELIGIBILITY:
Inclusion Criteria:

* Patients over the age of 65 who underwent surgery under spinal anesthesia due to hip fracture
* Volunteered to participate in the study

Exclusion Criteria:

* Patients who are under the age of 65
* Patients with known histories of dementia
* Patients with Alzheimer's disease
* Patients with central nervous system disease
* Patients who scored 15 or less according to the Mini Mental Status Test (MMSE)
* Patients who underwent surgery under general anesthesia
* Patients who refused to voluntarily participate in the study

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: Patients sedated with ketamine and dexmedetomidine during spinal anesthesia for hip fracture
Sampling Method: Probability Sample
Enrollment: 82 (Actual)
Dates: Start 2022-05-01 (Actual); Primary Completion 2022-12-31 (Actual); Study Completion 2022-12-31 (Actual)

PRIMARY OUTCOMES:
Mini-Mental Status Test | 6 months
  Evaluation of the effect of sedation with ketamine and dexmedetomidine on postoperative cognitive functions by Mini-Mental Status Test

SECONDARY OUTCOMES:
noninvasive mean arterial pressure | 6 months
  The effect of sedation on perioperative hemodynamics.
The heart rate | 6 months
  The effect of sedation on perioperative hemodynamics.

CONTACTS AND LOCATIONS:
Overall Officials: Derya A Yurtlu, M.D., Principal Investigator — Izmir Katip Celebi University Atatürk Training and Research Hospital
Locations (1):
- Izmir Katip Çelebi University Atatürk Training and Research Hospital, Izmir, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided